CLINICAL TRIAL: NCT04260360
Title: Phase 1 Trial Evaluating the Safety and Tolerability of NanoDoce® Intratumoral Injection in Subjects With Localized Renal Cell Carcinoma
Brief Title: Trial of NanoDoce Intratumoral Injection in Renal Cell Carcinoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Not initiated
Sponsor: NanOlogy, LLC (Industry)
Collaborators: US Biotest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NANODOCE-2018-01
Expanded Access: NCT04060628 (No longer available)
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Renal Cell Carcinoma; Kidney Cancer; Adenocarcinoma of Kidney; Adenocarcinoma, Renal; Renal Cell Cancer
Keywords: docetaxel
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Powders; Suspensions; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NanoDoce (Experimental): Intratumoral injection of NanoDoce (2.0 to 6.0 mg/mL) at a volume not to exceed 5.0 mL. NanoDoce will be administered on up to two occasions with at least 4 weeks between doses.
  Interventions: Drug: NanoDoce (sterile nanoparticulate docetaxel) Powder for Suspension

INTERVENTIONS:
Drug: NanoDoce (sterile nanoparticulate docetaxel) Powder for Suspension — NanoDoce is manufactured using a Precipitation with Compressed Antisolvent (PCA) technique that employs supercritical carbon dioxide and acetone to generate docetaxel nanoparticles within a well-characterized particle-size distribution. Prior to administration, the NanoDoce powder in vial is suspended with a sterile solution of Polysorbate 80 (0.0075% - 0.0375% (w/w))/Ethanol (0.06% - 0.3% (w/w)) in 0.9% Sodium Chloride for injection.
  Other Names: docetaxel

SUMMARY:
This study evaluates the use of NanoDoce injected directly into tumors in the kidney of people with renal cell carcinoma.

DETAILED DESCRIPTION:
NanoDoce is very small (submicron) particles of the chemotherapy drug, docetaxel, which is administered intravenously in a number of types of cancer. These submicron particles are injected directly into solid tumors to target cancer at the site of disease with less systemic exposure than intravenously administered chemotherapy. In this study, the submicron particle docetaxel will be injected directly into tumors in the kidney of people with renal cell carcinoma that is localized to (has not spread beyond) the kidney. All subjects in this study will receive NanoDoce and will be evaluated to see if NanoDoce is safe.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Age ≥18 years;
* Localized T1a renal cell carcinoma;
* Maximum tumor volume of 25.0 mL;
* Performance Status (ECOG) 0-2;
* Life expectancy of at least 6 months;
* Adequate marrow, liver, and renal function;

  * ANC ≥ 1.5 x 109/L
  * Hemoglobin ≥ 9.5 grams/dL
  * Platelets ≥ 75 x 109/L
  * Total bilirubin ≤ 1.5x institutional ULN
  * AST/ ALT ≤ 2.5x institutional ULN
  * Creatinine ≤ 1.5x institutional ULN
  * eGFR < 60 mL/min/1.73m2
* Adequate method of birth control.

Exclusion Criteria:

* Renal cyst;
* Multifocal or bilateral renal mass;
* Known hypersensitivity to any of the study drug or reconstitution components;
* Pregnant or breastfeeding female;
* Administration of an investigational product in a clinical trial within 3 months prior to consent;
* Investigator's opinion of subject's probable noncompliance or inability to understand the trial and/or give adequate informed consent;
* Known drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events | Day 1 to 180 days post-last NanoDoce injection
  Treatment emergent adverse events (including changes in laboratory assessments, physical examination findings, and vital signs)

SECONDARY OUTCOMES:
Concentration of docetaxel in the systemic circulation post-injection | Screening, Day 1, Day 2, Day 15, Day 27, Day 30, Day 31, Day 45, Month 2, Month 3, Month 4, Month 5, and 180 days post-last NanoDoce injection
  Pharmacokinetic samples will be obtained on the days of NanoDoce injection and other clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: Rose Marie Cavanna-Mast, RT, CCRA, Study Director — US Biotest, Inc.

IPD SHARING:
Plan to Share IPD: No